CLINICAL TRIAL: NCT03125733
Title: A Prospective International Multicenter Study on the Efficacy and Safety of Submucosal Tunneling Endoscopic Septum Division (STESD) for the Treatment of Zenker's Diverticulum
Brief Title: A New Treatment for Zenker's Diverticulum-submucosal Tunneling Endoscopic Septum Division
Acronym: STESD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Winthrop University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STESD for Zenker
Record Dates: First submitted 2017-04-16; First posted 2017-04-24 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Zenker Diverticulum
Keywords: Endoscopy, Digestive system; Natural orifice transluminal endoscopic surgery; Therapeutic; Complications
MeSH Terms: conditions — Zenker Diverticulum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- STESD (Experimental): Submucosal tunneling endoscopic septum division
  Interventions: Procedure: Submucosal tunneling endoscopic septum division

INTERVENTIONS:
Procedure: Submucosal tunneling endoscopic septum division — STESD includes 4 steps:
  1. Mucosal incision: submucosal injection of normal saline-indigo carmine solution is performed 2-3cm proximal to the diverticular septum and a 1.5-2cm longitudinal mucosal incision is made using the endoscopic knife.
  2. Submucosal tunneling: a submucosal tunnel is created using the same technique as applied by Peroral Endoscopic Myotomy (POEM) at both sides of the septum until 1-2cm distal to the bottom of the diverticulum.
  3. Septum Division: cricopharyngeal myotomy is performed longitudinally along the mid-line of the septum and ends in the normal esophageal muscle.
  4. Mucosal Closure: the mucosa incision, as well as any accidental mucosotomy if present, is closed with hemostatic clips.

SUMMARY:
Zenker's Diverticulum (ZD) is a sac-like outpouching of the lining of the esophageal wall at the upper esophagus. It is a rare disease typically seen in the middle-aged and older adults. Common symptoms of the disease include difficulties in swallowing (dysphagia), food reflux (regurgitation), unpleasant breath smells (halitosis) and couch, choking and hoarseness etc. (respiratory complications). Pills lodging in the sac and thus unable to take effect is also a common and yet often overlooked problem.

Traditional treatment for ZD included open resection done by head and neck surgeons and direct septum division done by ENT doctors. Septum division done by endoscopists is a new modality of treatment and so far has used the same approach as the ENT doctors-the wall between the sac and the normal esophageal lumen (the septum) is cut down directly so that food will not be held in the sac.

A cutting-edge endoscopic treatment for ZD is now emerging. In this approach, what we call submucosal tunneling endoscopic septum division (STESD), the wall is not cut directly, but inside a tunnel created by lifting the wallpaper (the mucosa lining the esophageal wall). After the muscle septum is completely cut, the mucosa is then sealed by clips, restoring integrity of the esophageal lining.

The advantage of STESD is twofold. First, the esophageal mucosa will be sealed after the operation, so that the chance of extravasation of luminal content with its relevant complications will be smaller. Second, under the protection of the tunnel, the endoscopist will be able to cut the septum completely down to its bottom, ensuring a more satisfactory symptom resolution. In short, our hypothesis is that treating Zenker's diverticulum by the tunneling endoscopic technique should be both safer and more effective than traditional methods.

DETAILED DESCRIPTION:
Patients with symptomatic Zenker's diverticulum are considered for STESD. The diagnosis is based on clinical presentation, barium swallow, EGD and a swallow test to rule out other possible disorders causing cervical dysphagia. A scoring system (Costamagna, GIE, 2016) is used to evaluate severity of the symptoms. Four symptoms are evaluated: 1) dysphagia, 2) regurgitation, 3) daytime respiratory symptoms and 4) nighttime respiratory symptoms. These are scored based on a solid food diet according to the symptom frequency calculated within 2 consecutive weeks: 0-never, 1-1day/ week, 2-2~4days/ week, 3-≥5 days/ week. Under EGD and barium swallow test, configuration of the diverticulum is documented in detail (Shou-Jiang Tang, Laryngoscope, 2008). Quality of life is assessed using the SF-36 form. The pre- and post-STESD symptom score, quality of life score, and diverticulum configuration are compared.

Adverse events are recorded and graded according to the system suggested by the ASGE workshop (Cotton, GIE, 2010).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Zenker's diverticulum by symptoms, esophagram and/ or EGD
* Symptomatic score≥2 in any of the symptoms or ≥3 in total
* Patients or legal surrogates willing and competent to give informed consent and to comply with follow up visits and tests

Exclusion Criteria:

* Patients with minimal symptoms (score ≤1 in all four symptoms and <3 in total)
* Presence of coagulopathy or pregnancy
* Patients who, in the investigator's opinion, are medically unstable or have a life expectancy of< 2 years, are unable to give informed consent or have poor compliance with follow-up, or whose risks of participating in the study outweigh the benefits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-06-14 (Estimated); Study Completion 2019-06-14 (Estimated)

PRIMARY OUTCOMES:
Short-term change of symptom score | 1 months after STESD
  Symptoms for Zenker's diverticulum are scored at follow-up visits and compared with pre-STESD value
Peri-operative adverse events | start of STESD to 30 days post-op
  Details and grading for any adverse event as defined by the ASGE lexicon are recorded during the peri-operative period

SECONDARY OUTCOMES:
Mid-term change of symptom score | 12 months after STESD
  Symptoms for Zenker's diverticulum are evaluated at follow-up visit and compared to pre-STESD value
Change of diverticulum size under EGD | 1 months after STESD
  ESD is done at follow-up visit and configuration of the diverticulum is compared to that pre-STESD
Change of diverticulum size under esophagram | 1 months after STESD
  Barium esophagram is done at follow-up visit and configuration of the diverticulum is compared to that pre-STESD
Call for other treatments, such as repeat myotomy | 12 months after STESD
  Call for any additional treatment for Zenker's diverticulum is recorded at follow-up visits

OTHER OUTCOMES:
Changes in quality of life score | Baseline and 12 months after STESD
  Patients' quality of life is recorded by using the SF-36 system

CONTACTS AND LOCATIONS:
Overall Officials: Ping-Hong Zhou, MD,PhD, Study Chair — Zhongshan Hospital, Fudan University, Shanghai, China; Stavros N Stavropoulos, MD, Study Director — NYU Winthrop Hospital, Mineola, NY, USA
Locations (2):
- NYU Winthrop Hospital, Mineola, New York, United States
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Costamagna G, Iacopini F, Bizzotto A, Familiari P, Tringali A, Perri V, Bella A. Prognostic variables for the clinical success of flexible endoscopic septotomy of Zenker's diverticulum. Gastrointest Endosc. 2016 Apr;83(4):765-73. doi: 10.1016/j.gie.2015.08.044. Epub 2015 Sep 3. PMID 26344886
- [Background] Tang SJ, Jazrawi SF, Chen E, Tang L, Myers LL. Flexible endoscopic clip-assisted Zenker's diverticulotomy: the first case series (with videos). Laryngoscope. 2008 Jul;118(7):1199-205. doi: 10.1097/MLG.0b013e31816e2eee. PMID 18401278
- [Background] Cotton PB, Eisen GM, Aabakken L, Baron TH, Hutter MM, Jacobson BC, Mergener K, Nemcek A Jr, Petersen BT, Petrini JL, Pike IM, Rabeneck L, Romagnuolo J, Vargo JJ. A lexicon for endoscopic adverse events: report of an ASGE workshop. Gastrointest Endosc. 2010 Mar;71(3):446-54. doi: 10.1016/j.gie.2009.10.027. No abstract available. PMID 20189503
- [Background] Gutschow CA, Hamoir M, Rombaux P, Otte JB, Goncette L, Collard JM. Management of pharyngoesophageal (Zenker's) diverticulum: which technique? Ann Thorac Surg. 2002 Nov;74(5):1677-82; discussion 1682-3. doi: 10.1016/s0003-4975(02)03931-0. PMID 12440629
- [Background] Ferreira LE, Simmons DT, Baron TH. Zenker's diverticula: pathophysiology, clinical presentation, and flexible endoscopic management. Dis Esophagus. 2008;21(1):1-8. doi: 10.1111/j.1442-2050.2007.00795.x. PMID 18197932
- [Background] Law R, Katzka DA, Baron TH. Zenker's Diverticulum. Clin Gastroenterol Hepatol. 2014 Nov;12(11):1773-82; quiz e111-2. doi: 10.1016/j.cgh.2013.09.016. Epub 2013 Sep 18. PMID 24055983
- [Background] Li QL, Chen WF, Zhang XC, Cai MY, Zhang YQ, Hu JW, He MJ, Yao LQ, Zhou PH, Xu MD. Submucosal Tunneling Endoscopic Septum Division: A Novel Technique for Treating Zenker's Diverticulum. Gastroenterology. 2016 Dec;151(6):1071-1074. doi: 10.1053/j.gastro.2016.08.064. Epub 2016 Sep 21. No abstract available. PMID 27664512
- [Background] Vigneswaran Y, Tanaka R, Gitelis M, Carbray J, Ujiki MB. Quality of life assessment after peroral endoscopic myotomy. Surg Endosc. 2015 May;29(5):1198-202. doi: 10.1007/s00464-014-3793-2. Epub 2014 Sep 24. PMID 25249144